CLINICAL TRIAL: NCT00412048
Title: Evaluation of fMRI-SAM in the Early Detection of Alzheimer's Disease.
Brief Title: Functional Magnetic Resonance Imaging - Synthetic Aperture Magnetometry (fMRI-SAM) and Alzheimer's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3659
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALZHEIMER DISEASE (Other)
  Interventions: Procedure: fMRI to detect MCI patients who will convert to Alzheimer's disease
- MOLD COGNITIVE IMPAIRMENT (Other)
  Interventions: Procedure: fMRI to detect MCI patients who will convert to Alzheimer's disease
- CONTROLS (Other)
  Interventions: Procedure: fMRI to detect MCI patients who will convert to Alzheimer's disease

INTERVENTIONS:
Procedure: fMRI to detect MCI patients who will convert to Alzheimer's disease — There is a fMRI to be realized in the 3 arms. No drug is administered

SUMMARY:
The aim of the protocol is to study the resting brain activation profile of 3 groups of people, using a new fMRI procedure, called fMRI-SAM. fMRI-SAM will be applied to 25 Alzheimer's disease (AD) patients, 25 patients suffering from amnestic - mild cognitive impairment (MCI) - a clinical picture which may be a prodromal form of AD - and 60 healthy controls. The first analysis of the data will search differences of brain activation profiles between the 3 groups. In the second step, the investigators will study the predictive value of fMRI-SAM to detect MCI patients who will later convert to AD.

ELIGIBILITY:
Inclusion criteria:

* Alzheimer's disease of mild to moderate severity (25 patients)
* Amnestic MCI patients (25 patients)
* 55-75 year-old patients

Exclusion criteria:

* Any other cause of dementia for AD patients
* Any stroke
* Any disease with a negative vital prognosis

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Comparing fMRI data between 3 groups of subjects: MCI, Alzheimer's disease and normal subjects | 1, 5 years

SECONDARY OUTCOMES:
Follow-up of MCI patients at 6, 12 and 18 months to detect a conversion to Alzheimer's disease | Prediction of Alzheimer's disease on fMRI data

CONTACTS AND LOCATIONS:
Overall Officials: Francois Sellal, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg